CLINICAL TRIAL: NCT00610129
Title: A Phase II Clinical and Translational Study of MK-0646 in Patients With Metastatic Neuroendocrine Tumors (NET)
Brief Title: Clinical and Translational Study of MK-0646 in Patients With Metastatic Neuroendocrine Tumors (NET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-162
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Neuroendocrine Tumors; Metastatic Neuroendocrine Tumors
Keywords: MK-0646
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — dalotuzumab

ARMS (1):
- 1 (Experimental): MK-0646
  Interventions: Drug: MK-0646

INTERVENTIONS:
Drug: MK-0646 — MK-0646 (20 mg/mL) in sterilized solution for IV infusion (12.7 mL to deliver 12.0 mL) will be used for a dose of 10 mg/kg IV weekly administered over 60 minutes.

SUMMARY:
The purpose of this study is to test a new drug for neuroendocrine tumors. We think that this new drug may help control your tumor.

MK-0646 is a monoclonal antibody. An antibody is a protein that is able to attach to specific target on cancer cells. This target helps the cancer cells grow and divide. By attaching to the target, it may stop the cancer cells from further growth and dividing. This study will help find out if MK-0646 is a helpful drug when taken in patients with neuroendocrine tumor.

This study is a phase 2 study. The purpose of a phase 2 study is to find out what effects, good and/or bad, MK-0646 has on metastatic neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic neuroendocrine tumors (NET)
* Patients must have histologically or cytologically confirmed well differentiated (low to intermediate grade) neuroendocrine tumors. High grade or poorly differentiated (i.e., large or small cell variant), Merkel cell, medullary carcinoma of the thyroid, and adrenal gland malignancies (including paragangliomas) are excluded from this study.
* Patient has at least one measurable lesion greater than or equal to 20 mm or greater than 10 mm on spiral CT.
* Patients who are on therapy with a somatostatin analogue are eligible for entry but must be on a stable dose for at least 3 months with no evidence of tumor shrinkage during that time period.
* Patient is male or female.
* Patient ≥ or equal to 18 years of age on the day of signing informed consent.
* Patient has performance status 0-2 on the ECOG Performance Scale.
* Patient has adequate organ function as indicated by the following laboratory values:
* Absolute Neutrophil Count (ANC) ≥ than or equal to 1,500/mcL
* platelets ≥ than or equal to 100,000/mcL
* Hemoglobin ≥ than or equal to 8 g/dL
* Serum Creatinine ≤ than or equal to 2 times the upper limit of normal (ULN)/ OR calculated CrCl ≥ than or equal to 60 mL/min (patients with creatinine levels ≥ than or equal to 2 times the ULN only). Patient may not be on dialysis
* Serum total bilirubin ≤ than or equal to 1.5 times the ULN
* AST (SGOT) and ALT (SGPT) ≤ than or equal to 5 times the ULN
* Prothrombin time (PT) Partial Thromboplastin time (PTT)
* ≤ than or equal to 1.2 times the ULN
* ≤than or equal to 1.2 times the ULN Creatinine clearance should be calculated by the Cockcroft-Gault method as follows:
* Male creatinine clearance = (140-age) x (weight in Kg)/(serum Cr x 72)
* Female creatinine clearance = ((140- age) x (weight in Kg)/(serum Cr x 72)) x 0.85
* Patient, or patient's legal representative, has voluntarily agreed to participate by giving written informed consent.
* Previous local therapy (e.g. chemoembolization or bland embolization) is allowed if completed > 6 weeks prior to study entry. For patients who received local therapy prior to study entry, there must be either documented growth of measurable disease within the embolization field or outside of the embolization field, or both, prior to study entry if the area of the embolization field was the only site of measurable disease.
* Previous chemotherapy, radiotherapy, and/or biologic therapy, including investigational agents, is/are allowed if completed > 4 weeks prior to study entry (>6 weeks if last regimen contained BCNU or mitomycin C, and > 6 weeks from last dose of radiation therapy or radiopharmaceutical.
* Patients must not have disease that is currently amenable to curative surgery. Prior surgery is allowed no less than 6 weeks prior to study entry.
* Patients with diabetes mellitus are eligible for study entry but must have controlled diabetes as defined by hemoglobin A1c <8.0% within 2 weeks of initiation of protocol therapy.

Exclusion Criteria:

* Patient has toxicities from prior therapies that have not resolved to grade 1 or grade 0.
* Patient has known CNS metastases and/or carcinomatous meningitis.
* Patient has known primary central nervous system tumor.
* Patient has a known hypersensitivity to the components of study drug (MK-0646) or its analogs that is not treatable by premedication with antihistamines and steroids.
* Patient has a condition, including but not limited to, serious active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or major psychiatric illness, which, in the opinion of the treating investigator, is likely to confound the results of the study, or makes participation not in the best interest of the patient.
* Patient has a history of a prior active malignancy within the past 5 years, with the exception of cervical intraepithelial neoplasia; basal cell carcinoma of the skin, adequately treated localized prostate carcinoma with PSA <1.0, or squamous cell carcinoma of the skin removed (or the more superficial keratoacanthoma).
* Patient has known psychiatric or substance abuse disorders that would, in the opinion of the treating investigator, interfere with cooperation with the requirements of the trial.
* Patient is breastfeeding or pregnant (this will requires a negative test within 72 hours of initiation of therapy), or expecting to conceive within the projected duration of the study.
* Patient is not using adequate contraception.
* Patient is known to be Human Immunodeficiency Virus (HIV)-positive.
* Patient has known active Hepatitis B or C.
* Patient is concurrently using growth hormone (GH), or growth hormone inhibitors.
* Patient has prior treatment with IGF-1R inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saltz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Metastatic Neuroendocrine Tumors: Translational Study of MK-0646 in Patients with Metastatic Neuroendocrine Tumors (NET)
Period: Overall Study
Arm/Group | Patients With Metastatic Neuroendocrine Tumors
Started | 28
Completed | 25
Not Completed | 3
Not completed — Not treated since patients ineligible | 3

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Metastatic Neuroendocrine Tumors
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: in patients with metastatic carcinoid tumors and in metastatic islet cell tumors (parallel cohorts) when treated with MK-0646 alone.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Patients With Metastatic Neuroendocrine Tumors
Number analyzed (Participants) | 25
participants
  Progression of Disease (POD) | 13
  Stable Disease (SD) | 12

ADVERSE EVENTS:
Arm/Group | Patients With Metastatic Neuroendocrine Tumors
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Metastatic Neuroendocrine Tumors (N=25)
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Nausea (General disorders) | 2 (2)
Pain - Abdomen NOS (General disorders) | 1 (1)
Pain - Neck (General disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Syncope (fainting) (General disorders) | 1 (1)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Metastatic Neuroendocrine Tumors (N=25)
ALT, SGPT (Blood and lymphatic system disorders) | 6 (6)
AST, SGOT (Blood and lymphatic system disorders) | 2 (2)
Albumin, low (hypoalbuminemia) (Blood and lymphatic system disorders) | 3 (3)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Renal and urinary disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (9)
Fever (in the absence of neutropenia) (General disorders) | 2 (2)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 14 (14)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Pain - Abdomen NOS (General disorders) | 4 (4)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes